CLINICAL TRIAL: NCT04591496
Title: The SmartFeeding4Kids, a Web-based Food Parenting Intervention to Promote Positive Feeding Practices and Healthy Diet in Preschool Children, Through Self-regulation and Behavior Change Techniques: a Randomized Control Trial
Brief Title: The SmartFeeding4Kids: Study of a New Web-based Food Parenting Intervention
Acronym: SF4K
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Lisbon (Other)
Collaborators: Faculdade de Psicologia, Universidade de Lisboa (Unknown); Centro de Investigação em Ciência Psicológica, Universidade de Lisboa (Unknown); FCiências.ID, Faculdade de Ciências, Universidade de Lisboa (Unknown); Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Luisa Barros, Full Professor, University of Lisbon
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PTDC/PSI-GER/30432/2017
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Parental Feeding Practices and Children's Healthy Diet
Keywords: Preschool child; Internet-based intervention; Parenting; Feeding behavior; Eating habits; Health education; Behavior change techniques; Random allocation
MeSH Terms: conditions — Feeding Behavior; Health Education

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of three groups in parallel for the duration of the study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SmartFeeding4Kids (Experimental): SmartFeeding4Kids: information about children's healthy diet and effective parental feeding practices, with a behavioral intervention (5 sessions plus 2 brief booster sessions online intervention)
  Interventions: Behavioral: Behavioral change intervention;; Behavioral: Health Education
- SmartFeeding4Kids Health (Active Comparator): Psychoeducational condition: information about children's healthy diet and effective parental feeding practices (5 sessions plus 2 brief booster sessions online intervention)
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Behavioral change intervention; — Behavioral change intervention: goal setting, regarding child's diet and parental feeding practices; self-monitoring, with observation and recording of the child's food intake and parental feeding practices; individualized feedback, based on preceding week monitoring and according to the defined objectives, regarding child's and parent's behaviors; modeling and direct suggestions by tailored parent figures; positive reinforcement associated to parents' accomplishment of the objectives; prompts, to remember the defined objectives and the main messages of the intervention.
  Arms: SmartFeeding4Kids
Behavioral: Health Education — Health education: provision of information about preschool children's nutrition guidelines, effective parental feeding practices, strategies to overcome food and feeding-related barriers, and steps to form healthy habits.

SUMMARY:
This research aims to develop and study the efficacy of a web-based brief intervention, Smart Feeding4Kids, to promote healthy dietary patterns in young children (2 to 6 years old) through changes in parents' feeding practices. The intervention is grounded on self-regulation and habit-formation models and combines the use of several effective behavioral methodologies. The multidisciplinary team integrates experienced researchers on parenting interventions, child nutrition, and the development of online applications to support personalized nutritional assessment and psychological interventions. The monitoring of the use of the platform and the knowledge about the predictors of efficacy, adherence, and involvement obtained in this project will offer professionals essential information to the development of future online interventions. The project will also contribute with knowledge concerning the most effective methodologies for changing parental feeding practices and collects unique information about the eating habits and practices of parents of Portuguese children.

The main hypotheses of the study:

1. parents who enrolled in behavior change and social support interventions will report significantly higher use of effective feeding practices (child's self-regulation intake practices, food availability, and accessibility practices) and significantly lower use of ineffective feeding practices (food control, restriction, and permissiveness feeding practices);
2. children whose parents enrolled in behavior change and social support interventions will have a significantly more frequent intake of vegetables and fruits intake, and significantly less frequent intake of sugar-sweetened foods and beverages;
3. positive changes in parental feeding practices will mediate children's food intake, with increased vegetables and fruits and decreased sugar-sweetened foods and beverages intake.

DETAILED DESCRIPTION:
A Randomized Control Trial with two groups (SmartFeeding4Kids, SmartFeeding4Kids Health) x 4 times (pre, post, 3-months, 6-month follow-up) repeated measures design will be used. Invitations to participate in the program will be made through flyers and social media messages. The invitation will show a link where parents can access detailed information about the program (study objectives, procedures, random allocation to one of the three conditions, data collected during the study). As this is a Randomized Control Trial study with repeated measurements, participants' identification must be recorded. The data relating to the parent's answers to evaluation protocols and self-monitoring, and time or interaction with the application/program, are associated with a personal account created by the participants at the beginning of the process. Consent protocol includes a paragraph that explains which data will be recorded and how it will be saved; parents must consent to researchers accessing this information. Only relevant information is collected. Data will be stored in a secure server. The team chose the server Amazon Web Services because is one of the most used services for hosting a website securely. Amazon Web Services delivers a mature set of services specifically designed for the unique security, compliance, privacy, and governance requirements of large organizations.

Once registered, parents are directed to the baseline assessment protocol. After the completion of the questionnaires and 24h food recalls, parents will be randomized and allocated to one of the two conditions through an automated web-based randomization program. For both conditions, parents will be invited to participate in five sessions plus two brief booster sessions. A new session is only accessible once parents have visualized the contents of the last session and performed the tasks proposed between sessions (for experimental conditions). Although the intervention is self-guided, each session is expected to be accomplished within an average of one week. At the end of the program, parents are redirected to fill the post-intervention assessment protocol; a similar procedure is performed after 3 and 6 months.

Cohen's f criteria will be used, with a small effect size of 0.15, an alpha equal to 0.05, and power of 0.80 for a two-group with four repeated measures design (with a moderate correlation pattern between time measurements of 0.35). The sample size needed is approximately 130 participants (i.e., 65 parents in each of the two-arm groups), but the total sample size was adjusted to account for a dropout rate of 50%. Therefore, the sample will be collected until 130 participants in each group (N = 260) finish the program. The proposed sample size will also be adequate for multilevel modeling with level-1 repeated measures nested within level-2 individuals, by assuring a minimum of 50 individuals required for level-2.

As mentioned before, the application does not allow participants to proceed to the sessions without completing all items of the baseline evaluation protocol, nor the participants have access to a new session if they do not complete the requested between-sessions records. As such, missing data will only be due to participant's dropout, during the intervention, or during the follow-up assessments completion. The researchers will use intention-to-treat principles: participants will be analyzed in the group in which they were allocated in the randomization process, independently of whether they had completed all measurement time points and/or the intervention. An evaluation of missing data mechanisms will be performed to inform which imputation strategy should be applied between multiple imputations (MI) and maximum likelihood estimation (FIML). Assuming the data are missing at random, a sensitivity analysis will be included, considering the whole samples vs. samples with complete data separately.

ELIGIBILITY:
Inclusion Criteria:

* Parent/caregiver of a 2 to 6 years old child, at baseline (if the parent has two children in the same age interval, the parent must choose the child that raises more concerns about their health habits, as reference)
* Have access to a mobile phone or computer/tablet with internet
* Be fluent in Portuguese
* Agree to participate in the study to accomplish the intervention in which they are allocated, the evaluation protocols, and the tasks required in each condition

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2021-07-13 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in the child's dietary intake reported by parents | Baseline, immediately after the intervention, 3 months after the intervention, 6 months after the intervention
  Child's dietary intake reported by parents: Child's dietary intake is evaluated through a 24h food recall, completed during 3 days (two weekdays and one weekend day). Data regarding the mean number of portions of vegetables, fruit, and sugar-sweetened foods and beverages registered on three days will be extracted from the database and analyzed separately as primary outcomes.
Changes from baseline in parental feeding practices | Baseline, immediately after the intervention, 3 months after the intervention, 6 months after the intervention
  Parental feeding practices: Parental feeding practices are evaluated through a self-reported questionnaire, Food Parenting Practices Questionnaire, with three subscales (Child's Intake Self-regulation Practices, Food Availability and Accessibility Practices, and Ineffective Control Practices) developed and adapted to the Portuguese population within this study. Parents answer to 40 items on a 5-point Likert scale (from Totally false to Totally true). Higher values on each subscale indicate a more frequent use of this type of parental feeding practices. The total mean score of each subscale ranged from 1 to 5.

SECONDARY OUTCOMES:
Changes from baseline in parental perceived barriers related to food and feeding | Baseline, immediately after the intervention, 3 months after the intervention, 6 months after the intervention
  Parental barriers are evaluated through a self-reported instrument, Parental Perception on Children's Healthy Feeding Barriers Questionnaire, developed and adapted to the Portuguese population within this study. The instrument has 30 items divided by 5 subscales (Child-related barriers, Parent-related barriers: vegetables & fruit, Parent-related barriers: added sugars, Context-related barriers, Cost-related barriers), answered on a 5-point Likert scale (from Totally false to Totally true). Higher values on each subscale indicate that a specific kind of parental barriers is more present. The total mean score of each subscale ranged from 1 to 5.
Changes from baseline in food parenting self-efficacy | Baseline, immediately after the intervention, 3 months after the intervention, 6 months after the intervention
  Parental self-efficacy is measured with a self-reported questionnaire, Parental Self-efficacy for Children's Healthy Diet Scale, previously developed by the team, with 4 items answered in a 5-point Likert scale (from No sure to Absolutely sure). Higher values on the scale correspond to higher parental self-efficacy. Score ranged from 1 to 5.
Changes from baseline in parental motivation to change | Baseline, immediately after the intervention, 3 months after the intervention, 6 months after the intervention
  Parental motivation to change is measured through a self-reported questionnaire with three items developed within this study. In each item, parents report their degree of importance, confidence and readiness to adhere and promote healthy changes in the child's diet and parental feeding practices, answering in a 10-point numerical scale (e.g., from Not important to Extremely important). Higher mean scores correspond to a higher degree of motivation to change (score ranged between 1 and 10).

OTHER OUTCOMES:
Perception of the child's weight | Baseline
  Parents are asked to subjectively rate their child's current weight, considering the child's age and height (underweight, average weight, overweight)
Concerns about the child's weight | Baseline
  Concerns about the child's weight are measured with four questions. The first question is about the parent's current concern about the child's weight. The other three items correspond to the Concern of Child Weight subscale of the Child Feeding Questionnaire - Revised (Birch et al., 2001) in its Portuguese version. The items are answered on a 5-point Likert scale (from No concern to Very concern). Higher values in the first item or in the subscale correspond to a higher degree of concerns about child's weight.
Child's BMI and percentile | Baseline, immediately after the intervention, 3 months after the intervention, 6 months after the intervention
  Children's weight and height measurements are assessed through parent's report. Child's BMI and percentile are calculated according to the World Health Organization Child Growth Standards.
Child's temperament | Baseline
  Parents are asked to read three sentences that describe the three temperament types and identify which better describe their child
Parent's BMI and percentile | Baseline
  Parent's weight and height measurements are assessed through their onw report. Parent's BMI and percentile are calculated according to the World Health Organization Standards.
Application usability | Immediately after the intervention
  To assess usability, we will use the System Usability Scale. It is a commonly used, validated 10-item questionnaire that asks users to rate a system on a 5-point Likert scale from '1= strongly disagree' to '5 = strongly agree'. Questions focus on the ease of use of the system and the integration of various functions within it.

CONTACTS AND LOCATIONS:
Overall Officials: Luisa Barros, Principal Investigator — University of Lisbon
Locations (1):
- Faculdade de Psicologia, Universidade de Lisboa, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Charneca S, Gomes AI, Branco D, Guerreiro T, Barros L, Sousa J. Intake of added sugar, fruits, vegetables, and legumes of Portuguese preschool children: Baseline data from SmartFeeding4Kids randomized controlled trial participants. Front Nutr. 2023 Mar 29;10:1150627. doi: 10.3389/fnut.2023.1150627. eCollection 2023. PMID 37063316
- [Derived] Gomes AI, Pereira AI, Guerreiro T, Branco D, Roberto MS, Pires A, Sousa J, Baranowski T, Barros L. SmartFeeding4Kids, an online self-guided parenting intervention to promote positive feeding practices and healthy diet in young children: study protocol for a randomized controlled trial. Trials. 2021 Dec 18;22(1):930. doi: 10.1186/s13063-021-05897-z. PMID 34922616